CLINICAL TRIAL: NCT00953602
Title: Long Time Metabolic Changes Induced by Genetically Modified Potatoes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Professor J. Spranger, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EA4/011/09
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Glucose Metabolism; Hormonal Changes; Satiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Genetically modified potato — Genetically modified potato

SUMMARY:
In this study the effects of genetically modified potatoes on the human metabolism will be observed. Healthy volunteers receive for one week muffins, produced with starch from a genetically modified potato or with a normal available starch, in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers

Exclusion Criteria:

* acute oder severe chronic diseases

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
glucose metabolism | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Charité, Dpt. of Endocrinology, Diabetes and Nutrition, Berlin, State of Berlin, Germany